CLINICAL TRIAL: NCT05192213
Title: Vitamin C, Hydrocortisone and Thiamine in Patients With Septic Shock: a Randomized Clinical Study (VITAMIN TRIAL)
Brief Title: Vitamin C, Hydrocortisone and Thiamine in Patients With Septic Shock
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In order to preserve the safety of the patients and prevent any harm from occurring, we opted to discontinue the study based on previous results (LOVIT study) published at 2022. Were recruited 71 than 1090 participants.
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: PROADI-SUS (Unknown); Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVAP-NG 1000; 07445119.9.1001.5461 (Other: Hospital Sirio-Libanês - Ethics Committee)
Record Dates: First submitted 2021-06-07; First posted 2022-01-14 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; vitamin C; thiamine; ICU
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Thiamine; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1,5 g of vitamin C every 6 hours + 200 mg of thiamine every 12 hours + 50 mg of hydrocortisone every 6 hours
  For 7 days or until patient's discharge/death
  Interventions: Drug: Vitamin C
- Control (Placebo Comparator): Placebo 1 for vitamin C every 6 hours + Placebo 2 for thiamine every 12 hours + 50 mg of hydrocortisone every 6 hours
  For 7 days or until patient's discharge/death
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin C — Patients will be allocated in a 1: 1 ratio to the treatment group, receiving intravenous Vitamin C (1.5 g every 6 hours), Thiamine (200 mg every 12 hours) and Hydrocortisone (50 mg every 6 hours) for 7 days
  Other Names: thiamine; hydrocortisone
  Arms: Intervention
Other: Placebo — Patients will receive 2 placebos (every 6 hours and every 12 hours) + Hydrocortisone (50 mg every 6 hours) for 7 days.
  Arms: Control

SUMMARY:
A great interest exists regarding substances with an immunomodulatory effect for sepsis patients. Recent data have shown that intravenous vitamin C, together with corticosteroids and thiamine, could prevent progressive organ dysfunction and reduce vasopressor use in patients with severe sepsis and septic shock. Its effect on mortality, on the other hand, is yet to be demonstrated. The Vitamins study aims to conclusively determine, through its prospective, multicentre and double-blinded design including 1090 patients, wether Vitamin C, Thiamine and Hydrocortisone in combination can reduce mortality in patients with septic shock.

DETAILED DESCRIPTION:
The global burden of sepsis is substantial with an estimated 15 to 19 million cases per year, most occurring in low-income countries. With recent advances in diagnosis and supportive treatment, the 28-day mortality from sepsis in high-income countries has decreased by about 25%; however, the mortality from septic shock still remains around 45%.

A large volume of experimental data has shown that both corticosteroids and intravenous vitamin C attenuate the release of pro-inflammatory mediators, reduce the endothelial lesion characteristic of sepsis (reducing endothelial permeability and improving microcirculatory flow), increase the release of endogenous catecholamines and improve vasopressor reaction. In animal models, these effects resulted in reduced organ damage and increased survival. However, its effect on critically ill humans is controvert. Results of a retrospective study brought that the early use of intravenous vitamin C, together with corticosteroids and thiamine, can prevent progressive organ dysfunction and can reduce mortality in patients with severe sepsis and septic shock.

For this reason, the investigators propose a randomized, controlled, multicentre (mcRCT), pragmatic and feasibility study to investigate whether Vitamin C (1.5g 6 / 6h), along with thiamine (200 mg, 12 / 12h) and hydrocortisone (50 mg 6 / 6h) for 7 days can reduce all-cause mortality within 28 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Sepsis of any background
* Vasopressor-dependent sepsis for at least 2 hours and vasopressor dose ≥ 0.25 µg / kg / min

Exclusion Criteria:

* Pregnancy;
* Requests for DNR (do not resuscitate) / DNI (do not intubate);
* Death is considered imminent or inevitable during this hospitalization and the attending physician, patient or substitute decision maker is not committed to active treatment;
* Patients with acute cerebral vascular event, acute coronary syndrome, active gastrointestinal bleeding, burn or trauma at admission;
* Patients with known HIV infection;
* Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency;
* Patients with septic shock transferred from another ICU or hospital with characteristics of septic shock for> 12 hours;
* Patients with septic shock characteristics for> 12 hours;
* Patients with a known history of oxalate nephropathy;
* Patients with short bowel syndrome or severe known fat malabsorption;
* Patients with acute beriberi disease;
* Patients with acute Wernicke's encephalopathy;
* Patients with known malaria;
* Patients with known or suspected scurvy;
* Patients with known or suspected Addison's disease;
* Patients with known Cushing's disease;
* Physician expects to prescribe or the patient has previously used (less than 15 days) systemic glucocorticoids for an indication other than septic shock (not including nebulized or inhaled corticosteroids), including the use of glucocorticoids for COVID-19;
* The patient is receiving treatment for systemic fungal infection or has documented Strongyloides infection at the time of randomization;
* Patient with known chronic iron overload due to iron storage and other diseases;
* Patient previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
28-day Mortality | 28 days
  Mortality by all causes at 28 days after randomization

SECONDARY OUTCOMES:
90-day Mortality | 90 days
  Mortality by all causes at 90 days after randomization
Duration of support | 28 days
  Duration of use of vasoactive drugs, mechanical ventilation and renal replacement therapy
Delta SOFA | 72 hours
  Change in total Sequential Organ Failure Assessment (SOFA) score, comparing SOFA score at 72 hours and SOFA score at randomisation. Range 0-24. Lower SOFA scores represent better outcome.
Quality of life assessment | 6 months
  Difference in quality of life assessment using the EQ-5D questionnaire, from EuroQol Group. The questionnaire will be applied during intensive care unit (ICU) stay and after 6 months. Range 0-1, with 0 and 1 corresponding to death and full health, respectively. This will be applied in 30% of research sample.

OTHER OUTCOMES:
Duration of hospital stay | Until hospital discharge or up to 90 days of randomisation
  Duration of hospital stay
Changes in Inflammatory Markers | Up to 96 hours of randomisation
  Analysis of procalcitonin and C-reactive protein collected at randomisation, after 48h and 96h after randomisation. This will be applied in 30% of research sample.
Incidence of Treatment-Emergent Adverse Events | 28 days
  Descriptive analysis of adverse events related to the study drugs, reported as incidence of the most recurrent events during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano CP Azevedo, PhD, Principal Investigator — Hospital Sirio-Libanês; Gisele Queiroz, MD, Principal Investigator — Hospitla Sirio-Libanês
Locations (12):
- Brazil (12):
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Hospital Otoclinica, Fortaleza, Ceará
  - Hospital Evangélico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital Clínica São Roque, Ipiaú, Estado de Bahia
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Passos, Passos, Minas Gerais
  - Hospital Universitário de Maringá, Maringá, Paraná
  - Hospital de Amor - Unidade Barretos, Barretos, São Paulo
  - Hospital SEPACO, São Paulo, São Paulo
  - Hospital Naval Marcílio Dias, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, São Paulo
  - Hospital São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
The study protocol and SAP are not submitted.

REFERENCES:
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518
- [Background] Vincent JL, Pereira AJ, Gleeson J, Backer D. Early management of sepsis. Clin Exp Emerg Med. 2014 Sep 30;1(1):3-7. doi: 10.15441/ceem.14.005. eCollection 2014 Sep. PMID 27752546
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Fujita I, Hirano J, Itoh N, Nakanishi T, Tanaka K. Dexamethasone induces sodium-dependant vitamin C transporter in a mouse osteoblastic cell line MC3T3-E1. Br J Nutr. 2001 Aug;86(2):145-9. doi: 10.1079/bjn2001406. PMID 11502226
- [Background] Marik PE. Critical illness-related corticosteroid insufficiency. Chest. 2009 Jan;135(1):181-193. doi: 10.1378/chest.08-1149. PMID 19136406
- [Background] he10 leading causes of death by country income group 2012. WHO factsheets. [http://www.who.int/mediacentre/factsheets/fs310/en/index1.html ]
- [Background] Sales Junior JA, David CM, Hatum R, Souza PC, Japiassu A, Pinheiro CT, Friedman G, Silva OB, Dias MD, Koterba E, Dias FS, Piras C, Luiz RR; Grupo de Estudo de Sepse do Fundo AMIB. [An epidemiological study of sepsis in Intensive Care Units: Sepsis Brazil study]. Rev Bras Ter Intensiva. 2006 Mar;18(1):9-17. Portuguese. PMID 25310321
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating sepsis. Cochrane Database Syst Rev. 2015 Dec 3;2015(12):CD002243. doi: 10.1002/14651858.CD002243.pub3. PMID 26633262
- [Background] Fujii T, Luethi N, Young PJ, Frei DR, Eastwood GM, French CJ, Deane AM, Shehabi Y, Hajjar LA, Oliveira G, Udy AA, Orford N, Edney SJ, Hunt AL, Judd HL, Bitker L, Cioccari L, Naorungroj T, Yanase F, Bates S, McGain F, Hudson EP, Al-Bassam W, Dwivedi DB, Peppin C, McCracken P, Orosz J, Bailey M, Bellomo R; VITAMINS Trial Investigators. Effect of Vitamin C, Hydrocortisone, and Thiamine vs Hydrocortisone Alone on Time Alive and Free of Vasopressor Support Among Patients With Septic Shock: The VITAMINS Randomized Clinical Trial. JAMA. 2020 Feb 4;323(5):423-431. doi: 10.1001/jama.2019.22176. PMID 31950979
- [Background] Hager DN, Hooper MH, Bernard GR, Busse LW, Ely EW, Fowler AA, Gaieski DF, Hall A, Hinson JS, Jackson JC, Kelen GD, Levine M, Lindsell CJ, Malone RE, McGlothlin A, Rothman RE, Viele K, Wright DW, Sevransky JE, Martin GS. The Vitamin C, Thiamine and Steroids in Sepsis (VICTAS) Protocol: a prospective, multi-center, double-blind, adaptive sample size, randomized, placebo-controlled, clinical trial. Trials. 2019 Apr 5;20(1):197. doi: 10.1186/s13063-019-3254-2. PMID 30953543
- [Background] Lindsell CJ, McGlothlin A, Nwosu S, Rice TW, Hall A, Bernard GR, Busse LW, Ely EW, Fowler AA, Gaieski DF, Hinson JS, Hooper MH, Jackson JC, Kelen GD, Levine M, Martin GS, Rothman RE, Sevransky JE, Viele K, Wright DW, Hager DN. Update to the Vitamin C, Thiamine and Steroids in Sepsis (VICTAS) protocol: statistical analysis plan for a prospective, multicenter, double-blind, adaptive sample size, randomized, placebo-controlled, clinical trial. Trials. 2019 Dec 4;20(1):670. doi: 10.1186/s13063-019-3775-8. PMID 31801567